CLINICAL TRIAL: NCT04351321
Title: A Multicenter, Randomized, Controlled Clinical Trial of the Safety of Totally Laparoscopic Versus Laparoscopy-Assisted Total Gastrectomy for Gastric Cancer.
Brief Title: The Safety of Totally Laparoscopic Versus Laparoscopy-Assisted Total Gastrectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLASS08
Record Dates: First submitted 2020-04-13; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Totally Laparoscopic Total Gastrectomy (Experimental): Totally laparoscopic total gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Totally Laparoscopic Total Gastrectomy
- Laparoscopy-Assisted Total Gastrectomy (Active Comparator): Laparoscopy-assisted total gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopy-Assisted Total Gastrectomy

INTERVENTIONS:
Procedure: Totally Laparoscopic Total Gastrectomy — Totally laparoscopic total gastrectomy will be performed in patients with gastric or esophagogastric junction adenocarcinoma of preoperative clinical stage I (T1N0M0, T1N1M0, T2N0M0) with D1+/D2 lymph node dissection.
  Arms: Totally Laparoscopic Total Gastrectomy
Procedure: Laparoscopy-Assisted Total Gastrectomy — Laparoscopy-Assisted Total Gastrectomy will be performed in patients with gastric or esophagogastric junction adenocarcinoma of preoperative clinical stage I (T1N0M0, T1N1M0, T2N0M0) with D1+/D2 lymph node dissection.
  Arms: Laparoscopy-Assisted Total Gastrectomy

SUMMARY:
To compare the short-term surgical safety and postoperative quality of life of totally laparoscopic versus laparoscopy-assisted total gastrectomy and to evaluate the superiority of totally laparoscopic total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years；
2. Primary lesion is diagnosed with endometrial biopsy as adenocarcinoma of the stomach or esophagogastric junction, including: papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), mixed adenocarcinoma, etc.；
3. Clinical stage cT1N0M0, cT1N1M0, cT2N0M0；
4. The gastric primary lesion is located in the body or fundus of stomach or the esophagogastric junction. It is expected that total gastrectomy with D1+/D2 lymph node dissection achieves R0 resection (multiple primary cancers are also applicable)；
5. BMI(Body Mass Index)<30 kg/m2；
6. No history of upper abdominal surgery (except for laparoscopic cholecystectomy)；
7. No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.；
8. Preoperative ECOG (Eastern Cooperative Oncology Group) performance status score 0 or 1；
9. Preoperative ASA (American Society of Anesthesiologists) scoring I-III；
10. Sufficient vital organ functions；
11. Signed informed consent.

Exclusion Criteria:

1. Preoperative examination indicates disease stage cStage II or above；
2. Women during pregnancy or lactation；
3. Suffer from other malignant tumors within 5 years；
4. Preoperative body temperature ≥ 38°C or complicated with infectious diseases requiring systemic treatment；
5. Severe mental illness；
6. Severe respiratory disease；
7. Severe liver and kidney dysfunction；
8. History of unstable angina or myocardial infarction within 6 months；
9. History of cerebral infarction or cerebral hemorrhage within 6 months；
10. Continuous application of glucocorticoid within 1 month (except for topical application)；
11. Accompanied by gastric cancer complications (bleeding, perforation, obstruction, etc.) ；
12. The patient has participated in or is participating in other clinical studies (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative morbidity | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complications are defined as the events observed within postoperative 30 days.

SECONDARY OUTCOMES:
Quality of life score | 3, 6 and 12 months
  Quality of life scores of the patients are evaluated based on EORTC C30 questionnaire at the 3rd, 6th and 12th months after operation.
Quality of life score | 3, 6 and 12 months
  Quality of life scores of the patients are evaluated based on STO22 questionnaire at the 3rd, 6th and 12th months after operation.
Overall incidence of postoperative morbidity | 12 months
  Refers to the incidence of overall postoperative complications observed during follow-up period.